CLINICAL TRIAL: NCT06562673
Title: Efficacy and Safety of Intra-arterial Cisplatin Plus Anti-angiogenesis Inhibitor Rh-endostatin (Endostar) Combined With Systematic Chemotherapy in Osteosarcoma
Brief Title: Intra-arterial Cisplatin Plus Rh-endostatin Combined With Systematic Chemotherapy in Osteosarcoma
Acronym: IACE-OS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hong-Tao Li, Principal Investigator, Shanghai 6th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-098-(1); 2024-098-(1) (Other: Approval Letter of Ethics Committee of Shanghai Sixth People's Hospital)
Record Dates: First submitted 2024-08-10; First posted 2024-08-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-08

CONDITIONS: Osteosarcoma; Bone Cancer
Keywords: osteosarcoma; intra-arterial; anti-angiogenesis inhibitor; endostatin; cisplatin
MeSH Terms: conditions — Osteosarcoma; Bone Neoplasms | interventions — endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IA cisplatin plus endostatin (Experimental): Intra-arterial cisplatin plus anti-angiogenesis inhibitor rh-endostatin (Endostar) combined with systematic chemotherapy
  Interventions: Drug: intra-arterial cisplatin plus anti-angiogenesis inhibitor rh-endostatin (Endostar)

INTERVENTIONS:
Drug: intra-arterial cisplatin plus anti-angiogenesis inhibitor rh-endostatin (Endostar) — After insertion of a catheter percutaneously by using the Seldinger technique through the brachial or femoral artery under local anesthesia, rh-endostatin was administered intra-arterially with dosage of 150 mg for a 6-h continuous infusion; then cisplatin was administered intra-arterially at 120 mg/m2 as a 6-h continuous infusion.
  Other Names: intra-arterial treatment

SUMMARY:
The goal of this clinical trial is to learn the efficacy and safety of intra-arterial cisplatin plus anti-angiogenesis inhibitor rh-endostatin (Endostar) combined with systematic chemotherapy in osteosarcoma. The main questions it aims to answer are:

* Is it safe when rh-endostatin and cisplatin are administered intra-arterially?
* Does intra-arterial cisplatin plus rh-endostatin increase the rate of tumor necrosis compared with traditional treatment?

Researchers will treat newly diagnosed osteosarcoma patients with systematic treatment and local treatment.

For systematic treatment, regular high-dose methotrexate and adriamycin will be administered intravenously.

For local treatment, rh-endostatin was administered intra-arterially with dosage of 150 mg for a 6-h continuous infusion; then cisplatin was administered intra-arterially at 120 mg/m2 as a 6-h continuous infusion.

Local treatment is conducted by insertion of a catheter percutaneously using the Seldinger technique through the brachial or femoral artery under local anesthesia.

Participants will:

• Receive local combined with systematic treatment once every 2-3 weeks for 2-4 cycles before surgery.

DETAILED DESCRIPTION:
Osteosarcoma (OS) is the most common bone cancer in children and young adolescents. Despite the emergence of new therapeutic modalities such as targeted therapy and immunotherapy, chemotherapy remains the standard treatment. The current standard treatment for osteosarcoma is the preoperative chemotherapy, surgery and postoperative chemotherapy. Preoperative chemotherapy (or neoadjuvant chemotherapy) and neoadjuvant chemotherapeutic agents include cisplatin, adriamycin, methotrexate. The use of preoperative chemotherapy has increased the 5-year survival rate from 20% to 60%-70%. Over the past 40 years, limited progress has been made in improving survival outcomes in patients with OS.

Transcatheter arterial infusion (TAI) is the direct infusion of drugs in the tumor blood supply artery, which can overcome the physiological barrier that some intravenous drug can not pass, thus significantly increasing the local drug concentration in the tumor and improving the therapeutic efficacy. Studies have shown that the combination of intravenous doxorubicin and intra-arterial cisplatin infusion before surgery resulted in a favorable histological response in 87% of enrolled patients, with a 10-year survival rate of 93% and an event-free survival rate of 86%.

Recombinant endostatin, an anti-angiogenic drug approved by the National Medical Products Administration of China in 2005 for the treatment of non-small cell lung cancer. In preclinical studies, synergistic antitumor efficacy was observed in an osteosarcoma mouse model with the addition of rh-endostatin to doxorubicin. In the clinical study of osteosarcoma, after comparing 58 patients with stage IIB osteosarcoma treated with chemotherapy combined with endostatin and 272 patients treated with chemotherapy alone, results show that the 5-year DMFS (distant metastasis-free survival) of the control group (61%) was significantly lower than that of the rh-endostatin group (79%) (P = 0.013). The 5-year OS of the control group (74%) was significantly lower than that of the rh-endostatin treatment group (87%) (P = 0.029). These results suggest that endostatin combined with chemotherapy for osteosarcoma significantly improves distant metastasis-free survival, with tolerable adverse effects, and is worthy of further clinical investigation.

Therefore, the investigators propose that arterial infusion of endostatin and cisplatin combined with systematic therapy might improve the treatment efficacy in preoperative course.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of osteosarcoma patients aged 12-40 years old;
2. Accept to receive treatment with neoadjuvant chemotherapy regimen and completing the standard treatment course; Voluntary informed consent, joining the study with good compliance.
3. Have detailed medical data (such as medical history data, laboratory reports of blood routine and liver and kidney functions, pathology reports, etc.), and complete records of postoperative follow-up.

Exclusion Criteria:

1. Combined history of acute injury, infection and surgery in the last 3 months;
2. Those with severe liver and kidney function abnormalities;
3. Those who are using anti-inflammatory drugs;
4. Pre-existing hematologic diseases before treatment;
5. Combined with other malignant tumors;
6. Diagnosed with autoimmune disease or using steroid drugs for more than 1 month before treatment;
7. Suffering from mental illness or cognitive dysfunction.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From enrollment to the end of treatment at 1-month
  Safety analysis (adverse events) according to CTCAE 5.0
Incidence of tumor response | From enrollment to the end of treatment at 1 month
  according to tumor cell necrosis rate (TCNR) of tumor tissue sample after surgery.

SECONDARY OUTCOMES:
Microvessel density | From enrollment to the end of treatment at 1 month
  the measurement of microvessel density (MVD) detected in tumor tissue sample after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Tao Li, Dr., Principal Investigator — Shanghai Jiao Tong University School of Medicine, Shanghai Sixth People's Hospital
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai Sixth People's Hospital,, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
only IPD used in the results publication

REFERENCES:
- [Background] Xu H, Huang Z, Li Y, Zhang Q, Hao L, Niu X. Perioperative rh-endostatin with chemotherapy improves the survival of conventional osteosarcoma patients: a prospective non-randomized controlled study. Cancer Biol Med. 2019 Feb;16(1):166-172. doi: 10.20892/j.issn.2095-3941.2018.0315. PMID 31119057
- [Background] Shaikh R, Munoz FG. Endovascular approaches in pediatric interventional oncology. CVIR Endovasc. 2021 Jan 2;4(1):2. doi: 10.1186/s42155-020-00190-7. PMID 33387076
- [Background] Xie L, Xu J, Dong S, Gao J, Tang X, Yan T, Yang R, Guo W. Gain and loss from transcatheter intra-arterial limb infusion of cisplatin for extremity osteosarcoma: a retrospective study of 99 cases in the past six years. Cancer Manag Res. 2019 Jul 30;11:7183-7195. doi: 10.2147/CMAR.S214604. eCollection 2019. PMID 31447583
- [Background] Avritscher R, Javadi S. Transcatheter intra-arterial limb infusion for extremity osteosarcoma: technical considerations and outcomes. Tech Vasc Interv Radiol. 2011 Sep;14(3):124-8. doi: 10.1053/j.tvir.2011.02.004. PMID 21767779
- [Background] Zhang HJ, Yang JJ, Lu JP, Lai CJ, Sheng J, Li YX, Hao Q, Zhang SM, Gupta S. Use of intra-arterial chemotherapy and embolization before limb salvage surgery for osteosarcoma of the lower extremity. Cardiovasc Intervent Radiol. 2009 Jul;32(4):672-8. doi: 10.1007/s00270-009-9546-2. Epub 2009 Mar 19. PMID 19296158
- [Background] Wilkins RM, Cullen JW, Camozzi AB, Jamroz BA, Odom L. Improved survival in primary nonmetastatic pediatric osteosarcoma of the extremity. Clin Orthop Relat Res. 2005 Sep;438:128-36. doi: 10.1097/01.blo.0000179736.10871.76. PMID 16131881
- [Background] Wilkins RM, Cullen JW, Odom L, Jamroz BA, Cullen PM, Fink K, Peck SD, Stevens SL, Kelly CM, Camozzi AB. Superior survival in treatment of primary nonmetastatic pediatric osteosarcoma of the extremity. Ann Surg Oncol. 2003 Jun;10(5):498-507. doi: 10.1245/aso.2003.03.061. PMID 12794015
- [Background] Rao BN, Rodriguez-Galindo C. Intra-arterial cisplatin in osteosarcoma: same question, different answer. Ann Surg Oncol. 2003 Jun;10(5):481-3. doi: 10.1245/aso.2003.04.903. No abstract available. PMID 12794009
- [Background] Wanebo HJ, Temple WJ, Popp MB, Constable W, Aron B, Cunningham SL. Preoperative regional therapy for extremity sarcoma. A tricenter update. Cancer. 1995 May 1;75(9):2299-306. doi: 10.1002/1097-0142(19950501)75:93.0.co;2-y. PMID 7712441
- [Background] Bielack SS, Bieling P, Erttmann R, Winkler K. Intraarterial chemotherapy for osteosarcoma: does the result really justify the effort? Cancer Treat Res. 1993;62:85-92. doi: 10.1007/978-1-4615-3518-8_12. PMID 8096763